CLINICAL TRIAL: NCT01100970
Title: Cortisol Levels in Infants Born by C-section - A Comparison of Using an Electric Unipolar Needle and Electric Bipolar Needle
Brief Title: Cortisol Levels in Infants Born by C-section - Electric Unipolar Needle Versus Electric Bipolar Needle
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: David Mankuta, MD, Hadassah Ein-Kerem - obstetrics and gynecology
Other Study IDs: 0008-10HMO-CTIL
Record Dates: First submitted 2010-04-08; First posted 2010-04-09 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2010-02

CONDITIONS: Delivery
Keywords: Caesarean section; cortisol; stress; unipolar electric needle; bipolar electric needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bouth umbilical Blood samples and saliva samples will be kept in a -20C freezer utill assayed.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Unipolar electric needle
- Bipolar electric needle
- Control: Infants who were born in a vaginal birth

SUMMARY:
The purpose of this study is to determine whether there is a difference between cortisol levels in fetal blood of babies who were born while using a unipolar needle opposite to using a bipolar needle, and compared to the control group (infants who were born in a vaginal birth).

DETAILED DESCRIPTION:
Today, on Caesarean section, there's a widely usage of electric unipolar needle for cutting tissue and / or bipolar needle to burn blood vessels. These Needles use an electric current flow for cutting the tissue. When using unipolar needle there's a transfer of the electric current through the mother's body and through the amniotic fluid , while when using bipolar needle the current goes back through the needle directly the generator so that the flow does not transfer to the amniotic fluid and fetus.

Despite the growing usage of electric needles, there is no literature information about the extent of electrical current that is transferred to the fetus during cutting, hence, no information about stress level felt by the baby as a result of electrical current exposure.

The purpose of this experiment is testing the possibility that there is a difference between cortisol levels in fetal blood of babies who were born while using a unipolar needle opposite to using a bipolar needle, and compared to the control group (infants who were born in a vaginal birth).

Also, we want to check whether there is correlation between maternal cortisol levels and newborn cortisol levels (whether motherly cortisol levels affects newborn cortisol levels).

To assess cortisol at birth, blood will be taken from the umbilical vein following clamping of the cord after birth. Saliva-based cortisol will be collected from mothers.

Other measures which will be taken are: week of birth, newborns weight, Apgar score 5 minutes after birth, mother's age and the indication for cesarean section.

Then we will compare the two experimental groups, as well as compare the two groups, to the control group, and see whether there is a statistically significant difference between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women, without significant background and/or chronic diseases.
2. Women who did not experienced illnesses that may pass to the fetus during pregnancy, or any other medical complication related to pregnancy.
3. All indications for C-section are medical indications.
4. Male newborn, week 37-42 of pregnant.
5. Without any evidence of stress event suffered by the mother or fetus during pregnancy or at birth.

Exclusion Criteria:

1. Women over 45 years of age, or under the age of 20.
2. Women with significant background and/or chronic diseases.
3. Women who experienced medical complications during pregnancy.
4. C-section indication are urgent due to mother/fetus distress.
5. Female newborn, or a male newborn who wasn't born during week37-42 of pregnancy.
6. Evidence of a stress event suffered by the mother and/or fetus during pregnancy or at birth.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women who needs c-section.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Mankuta, MD, Principal Investigator — Hadassah University Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Gitau R, Menson E, Pickles V, Fisk NM, Glover V, MacLachlan N. Umbilical cortisol levels as an indicator of the fetal stress response to assisted vaginal delivery. Eur J Obstet Gynecol Reprod Biol. 2001 Sep;98(1):14-7. doi: 10.1016/s0301-2115(01)00298-6. PMID 11516793